CLINICAL TRIAL: NCT06340438
Title: Investigation of the Neurophysiological and Psychological Aspects of Itch
Brief Title: Investigate the Relationship Between Catastrophizing and the Perception of Itch Intensity in Healthy Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Associate Professor, Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20240004 3rd subproject
Record Dates: First submitted 2024-03-19; First posted 2024-04-01 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Histamine; Cowhage
MeSH Terms: interventions — Histamine

STUDY DESIGN:
Intervention Model Description: The participants will randomly receive applications of cowhage and histamine.
Who Masked: Participant
Masking Description: Participant will be blinded about application of pruritogens.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Histamine application (Other): In the first session, the subjects will fill some questionnaires. After that, a squared area of 4x4 cm will be selected at the center of each middle forearm of the subject and cowage or histamine will be applied for 10 minutes, during which the pain/itch following the cowhage/histamine application will be monitored with a VAS scale. After the itch-induction, the subjects will fill in other questionnaire. In second session, the subjects will fill some questionnaires. After that, a squared area of 4x4 cm will be selected at the center of each middle forearm of the subject and cowage or histamine will be applied for 10 minutes, during which the pain/itch following the cowhage/histamine application will be monitored with a VAS scale. After the itch-induction, the subjects will fill out other questionnaires. The order will be randomized, so if the subjects were given the cowhage in the first session, they will receive the histamine application in the second session, and vice versa.
  Interventions: Other: Histamine
- Cowhage application (Other): In the first session, the subjects will fill some questionnaires. After that, a squared area of 4x4 cm will be selected at the center of each middle forearm of the subject and cowage or histamine will be applied for 10 minutes, during which the pain/itch following the cowhage/histamine application will be monitored with a VAS scale. After the itch-induction, the subjects will fill in other questionnaire. In second session, the subjects will fill some questionnaires. After that, a squared area of 4x4 cm will be selected at the center of each middle forearm of the subject and cowage or histamine will be applied for 10 minutes, during which the pain/itch following the cowhage/histamine application will be monitored with a VAS scale. After the itch-induction, the subjects will fill out other questionnaires. The order will be randomized, so if the subjects were given the cowhage in the first session, they will receive the histamine application in the second session, and vice versa.
  Interventions: Other: Cowhage

INTERVENTIONS:
Other: Histamine — Histaminergic itch will be evoked by a 1% histamine solution. A droplet of histamine solution will be placed on the predetermined area on the forearm, and the SPT lancet will be pierced through the histamine with 120 g of pressure for 1-2 seconds.
  Arms: Histamine application
Other: Cowhage — 25 spicules will be inserted in the center of the predefined skin area on the mandibular area. The spicules will be gently rubbed for 15-20 seconds in circular motion to facilitate epidermal penetration.
  Arms: Cowhage application

SUMMARY:
This project aims to investigate the relationship between different dimensions of catastrophizing (rumination, magnification, and helplessness) as well as some specific personality traits related to catastrophizing tendencies like anxiety sensitivity and fear sensitivity in the modulation of itch and pain intensities in an experimental setting.

DETAILED DESCRIPTION:
Chronic itch severely affects the quality of life of patients by interfering with vital functions such as sleep, attention, and sexual activity, with an elevated expression of cognitive and emotional factors such as itch catastrophizing, worrying, as well as personality characteristics such as the predisposition to anxiety, depression, and suicidal thoughts that play an important role in the development, modification, and maintenance of itch. Moreover, chronic itch represents a significant socioeconomic burden due to a prevalence of around 10% in combination with largely suboptimal treatment since limited evidence has been found for the effectiveness of pharmaceutical interventions. The hypothesis of this project is that since it is well documented that the relationship between catastrophizing and pain and that itch and pain share many similarities, investigators can assume the existence of a similar connection between catastrophizing and itching.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids, or other addictive drugs
* Previous or current history of neurological (e.g. neuropathy), immunological (e.g. asthma, immune deficiencies, arthritis), musculoskeletal (e.g. muscular pain in the upper extremities,), cardiac disorder, or mental illnesses that may affect the results
* Lack of ability to cooperate
* Current use of medications that may affect the trial such as antihistamines, antipsychotics, and pain killers, as well as systemic or topical steroids
* Skin diseases (e.g. atopic dermatitis, pruritus nodularis, eczema, psoriasis)
* Moles, scars, or tattoos in the area to be treated or tested.
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain
* Participation in other trials within one week of study entry (four weeks in the case of pharmaceutical trials)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-04-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Reinforcement Sensitivity Theory - Personality Questionnaire (RST-PQ). | Baseline 1st session
  The Reinforcement Sensitivity Theory - Personality Questionnaire contains the following subscales: the Fight-Flight-Freeze System (FFFS, 10 items); the Behavioral Inhibition System (BIS, 23 items); and the Behavioral Approach System (BAS, 32 items). In total, 65 items have to be answered on a 4-point Likert-type scale ranging from 1 (not at all) to 4 (Highly).
The Pittsburg Sleep Quality Index (PSQI) | Baseline 1st session
  The PSQI consists of 19 items generating seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The seven component scores can be summarized in a global score ranging from zero to 21 with higher scores reflecting a worse overall quality of sleep.
Depression, Anxiety, Stress Scale (DASS-21) | Baseline 1st session
  The questionnaire measures the magnitude of depression, anxiety, and stress. Each of these three subscales consists of 7 questions answered using a 0-3 Likert scale, with 0 meaning "it did not apply to me", and 3 meaning "it applied to me very much"
Positive And Negative Affect Schedule (PANAS) | Baseline 1st session
  PANAS measures positive and negative affect dimensions. Positive affects (PA) are defined as "the extent to which a person feels active, enthusiastic, and alert". Negative affect (NA) is a condition of "general distress and unpleasable engagement".
Pain Catastrophizing Scale (PCS). | 10 minutes after every itch induction on 1st session
  The PCS assesses negative and exaggerated coping concerning anticipated or experienced painful stimuli. Thirteen items have to be answered on a 5-point Likert-type scale ranging from 0 (Not at all) to 4 (all the time).
Itch Catastrophizing Scale (ICS). | 10 minutes after every itch induction on 1st session
  The ICS assesses negative and exaggerated coping concerning anticipated or experienced itchy stimuli. Thirteen items have to be answered on a 5-point Likert-type scale ranging from 0 (Not at all) to 4 (all the time).
Learned Helplessness Scale (LHS) | 10 minutes after every itch induction on 1st session
  The questionnaire consists of 20 items, and the participant's response to each item is rated on a 4-point Likert scale ranging from strongly agree (1) to strongly disagree (4).
Positive And Negative Affect Schedule (PANAS) | 10 minutes after every itch induction on 1st session
  PANAS measures positive and negative affect dimensions. Positive affects (PA) are defined as "the extent to which a person feels active, enthusiastic, and alert". Negative affect (NA) is a condition of "general distress and unpleasable engagement".
Depression, Anxiety, Stress Scale (DASS-21) | Baseline 2nd session (3 days after 1st session)
  The questionnaire measures the magnitude of depression, anxiety, and stress. Each of these three subscales consists of 7 questions answered using a 0-3 Likert scale, with 0 meaning "it did not apply to me", and 3 meaning "it applied to me very much"
Positive And Negative Affect Schedule (PANAS) | Baseline 2nd session (3 days after 1st session)
  PANAS measures positive and negative affect dimensions. Positive affects (PA) are defined as "the extent to which a person feels active, enthusiastic, and alert". Negative affect (NA) is a condition of "general distress and unpleasable engagement"
Pain Catastrophizing Scale (PCS). | 10 minutes after every itch induction on 2nd session (3 days after 1st session)
  The PCS assesses negative and exaggerated coping concerning anticipated or experienced painful stimuli. Thirteen items have to be answered on a 5-point Likert-type scale.
Itch Catastrophizing Scale (ICS). | 10 minutes after every itch induction on 2nd session (3 days after 1st session)
  The ICS assesses negative and exaggerated coping concerning anticipated or experienced itchy stimuli. Thirteen items have to be answered on a 5-point Likert-type scale.
Learned Helplessness Scale (LHS) | 10 minutes after every itch induction on 2nd session (3 days after 1st session)
  The questionnaire consists of 20 items, and the participant's response to each item is rated on a 4-point Likert scale ranging from strongly agree (1) to strongly disagree (4).
Positive And Negative Affect Schedule (PANAS) | 10 minutes after every itch induction on 2nd session (3 days after 1st session)
  PANAS measures positive and negative affect dimensions. Positive affects (PA) are defined as "the extent to which a person feels active, enthusiastic, and alert". Negative affect (NA) is a condition of "general distress and unpleasable engagement"

SECONDARY OUTCOMES:
Assessment of itch | 1 minute after every itch inductions
  Immediately following the itch provocations, participants will be instructed to rate the itch intensity for 10 minutes using a digital visual analogue scale (VAS; eVAS Software: Aalborg, University, Denmark), on a tablet. The scale will be measured from 0 to 100, where 0 represents 'no itch' and 100 'worst itch imaginable'.
Assessment of pain | 1 minute after every itch inductions
  Immediately following the itch provocations, participants will be instructed to rate the pain intensity for 10 minutes using a digital visual analogue scale (VAS; eVAS Software: Aalborg, University, Denmark), on a tablet. The scale will be measured from 0 to 100, where 0 represents 'no pain' and 100 'worst pain imaginable'.

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, Denmark